CLINICAL TRIAL: NCT02525783
Title: Aequalis Pyrocarbon Humeral Head IDE Study
Brief Title: Aequalis Pyrocarbon IDE; Replacing the Humeral Head in Hemi-Arthroplasty
Acronym: PYC
Status: Completed | Type: Interventional
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15A-T-PYC-R
Record Dates: First submitted 2015-08-14; First posted 2015-08-17 (Estimated); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis; Avascular Necrosis; Traumatic Arthritis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Hemi Shoulder Arthroplasty (Experimental): Hemi Shoulder Arthroplasty using the Aequalis Pyrocarbon Humeral Head
  Interventions: Device: Aequalis Pyrocarbon Humeral Head

INTERVENTIONS:
Device: Aequalis Pyrocarbon Humeral Head — Hemi Shoulder Arthroplasty

SUMMARY:
The purpose of this study is to demonstrate safety and effectiveness of the Aequalis Pyrocarbon Humeral Head in hemiarthroplasty at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject 22 years or older.
* Scapula and proximal humerus must have reached skeletal maturity.
* Clinical indication for hemiarthroplasty due to primary diagnosis of arthritis or avascular necrosis. Primary arthritis for this study includes osteoarthritis with pain and/or post-traumatic arthritis.
* Willing and able to comply with the protocol.
* Willing and able to sign the informed consent formed (or the Legally Authorized Representative will sign for the subject).

Exclusion Criteria:

* Active local or systemic infection, sepsis, or osteomyelitis.
* In the opinion of the clinician, there is insufficient bone stock to support implants in the humeral metaphysis or poor bone quality.
* In the opinion of the clinician, there is insufficient bone stock or excessive deformation of the native glenoid to allow normal functioning of the glenohumeral joint.
* In the clinician's opinion, the subject is unwilling or unable to be compliant with the recommendations of the healthcare professional.
* Metabolism disorders that could compromise bone formation, or Osteomalacia.
* Infection at or near the implant site, distant foci of infections that could spread to the site of the implant, or systemic infection.
* Rapid destruction of the joint, marked bone loss, or bone resorption apparent on X-ray.
* Known allergy or suspected allergy to implant materials.
* Female subjects who are pregnant or planning to become pregnant within the study period.
* Medical conditions or balance impairments that could lead to falls. Prior arthroplasty or prior failed rotator cuff repair on the affected shoulder; (successful rotator cuff surgery may be included).
* A rotator cuff that is not intact and cannot be reconstructed. Subjects with a massive rotator cuff tear (>5cm) will be excluded.
* Nonfunctional deltoid muscle.
* Neuromuscular compromise condition of the shoulder (e.g., neuropathic joints or brachial plexus injury with a flail shoulder joint).
* Known active metastatic or neoplastic diseases, Paget's disease, or Charcot's disease.
* Currently, within the last 6 months, or planning to be on chemotherapy or radiation.
* Known alcohol or drug abuse as defined by DSM-5.
* Taking greater than 5mg/day corticosteroids (e.g. prednisone) excluding inhalers, within 3 months prior to surgery.
* Currently enrolled in any clinical research study that might interfere with the current study endpoints.
* Known history of renal or hepatic disease/insufficiency.
* Anatomy cannot be replicated using current available system sizes.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2015-12; Primary Completion 2019-07-19 (Actual); Study Completion 2022-10-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers. Only aggregate data will be shared with the researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Tornier Pyrocarbon Humeral Head: The Tornier Pyrocarbon Humeral Head associated with the Tornier Flex stem. The Aequalis Pyrocarbon Humeral Head shoulder prosthesis, combined with the Aequalis Ascend Flex stem, is to be used only in patients with an intact or reconstructable rotator cuff and if the native glenoid surface is intact or sufficient, where they are intended to increase mobility, stability, and relieve pain. This is a hemiarthroplasty procedure.
Period: Overall Study
Arm/Group | Tornier Pyrocarbon Humeral Head
Started | 157
Completed | 147
Not Completed | 10
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Arm/Group | Tornier Pyrocarbon Humeral Head
Number analyzed (Participants) | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 124
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Constant Score [Mean (Standard Deviation); unit: units on a scale] — Constant Score: In this score, 35 points are allocated for subjective assessments of pain and activities of daily living and 65 points are available for objective measures of range of movement and shoulder strength. A young healthy patient can therefore have a maximum score of 100 points. The minimum score is 0 points. A higher value represents a better outcome.
  * Average of 2 pain scores (15 points max)
  * Sum of 4 activities of daily living questions (20 points max)
  * Sum of 4 ROM measure (40 points max)
  * Power score (25 points max)
  units on a scale | 42.6 (15.0)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Patient Success at 24 Months.
Description: A subject is a success at 24 months if:
  * Their change in Constant score is greater than or equal to 17 and
  * They did not have revision surgery; and
  * There is no radiographic evidence of system disassembly or fracture, and
  * They did not have a system-related serious adverse event.
Time Frame: 24 Months
Population: This number of participants is 146 as 10 patients were lost to follow-up (were not seen at 24 months) and one patient did not have a baseline Constant Score.
Measure: Count of Participants; unit: Participants
Arm/Group | Tornier Pyrocarbon Humeral Head
Number analyzed (Participants) | 146
Participants | 120

2. Secondary Outcome: Constant Score
Description: Constant Score: In this score, 35 points are allocated for subjective assessments of pain and activities of daily living and 65 points are available for objective measures of range of movement and shoulder strength. A young healthy patient can therefore have a maximum score of 100 points. The minimum score is 0 points. The range of the score is 0-100 for both the Constant Score and the adjusted Constant score. A higher value represents a better outcome.
  Average of 2 pain scores (15 points max) Sum of 4 activities of daily living questions (20 points max) Sum of 4 ROM measure (40 points max) Power score (25 points max)
  Change in Constant Score and Adjusted Constant Score at 24 months compared to baseline is presented along with absolute values.
Time Frame: 24 Months
Population: 143 were analyzed as 10 patients were lost to follow-up, one patient did not have a baseline Constant Score, and three patients were revised prior to a 24-month visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tornier Pyrocarbon Humeral Head
Number analyzed (Participants) | 143
units on a scale
  Constant Score Increase (change in score) | 34.3 (17.8)
  Adjusted Constant Score Increase (change in score) | 39.5 (20.5)
  Constant Score (Absolute value) | 78.1 (16.4)

3. Secondary Outcome: American Shoulder and Elbow Surgeons (ASES) Score
Description: American Shoulder and Elbow Surgeons Standardized Shoulder Assessment. The original ASES consists of 2 portions, a medical professional assessment section and a patient self-report section. The patient self-report section utilized in this study is a condition specific scale intended to measure functional limitations and pain of the shoulder. The assessment takes approximately 5 minutes to complete and consists of 2 dimensions: pain and activities of daily living. The pain score is calculated from the single pain question and the function score from the sum of the 10 questions addressing function. The pain score and function composite score are weighted equally (50 points each) and combined for a total score out of a possible 100 points. The minimum score is 0 and the maximum score is 100. A higher value represents a better outcome.
  Change in American Shoulder and Elbow Surgeons (ASES) Score at 24 months compared to baseline are presented.
Time Frame: 24 Months
Population: ASES Increase reported. 144 were analyzed as 10 patients were lost to follow-up (no 24-month visit) and three patients were revised prior to the 24-month visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tornier Pyrocarbon Humeral Head
Number analyzed (Participants) | 144
units on a scale
  ASES Score Increase (Change from Baseline) | 43.4 (21.7)
  ASES Score (Absolute value) | 87.5 (17.5)

4. Secondary Outcome: Single Assessment Numeric Evaluation (SANE)
Description: The SANE rating is determined by the subject's written response to the following question "How would you rate your shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?"
  Change in Single Assessment Numeric Evaluation (SANE) at 24 months compared to baseline
Time Frame: 24 Months
Population: SANE score increase reported. 144 were analyzed as 10 patients were lost to follow-up and three patients were revised prior to 24-month visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tornier Pyrocarbon Humeral Head
Number analyzed (Participants) | 144
score on a scale
  SANE Score Increase (Change from baseline) | 49.5 (26)
  SANE Score (Absolute Value) | 85.4 (19.1)

5. Secondary Outcome: EQ-5D Index
Description: EQ-5D: a standardized instrument for use as a measure of health outcome. It is cognitively simple, takes only a few minutes to complete, and provides a simple descriptive profile as well as a single index value for health status. Scale 0 to 1; 1 (representing full health) to 0 (representing dead).
  Change in EQ-5D score at 24 months compared to baseline
Time Frame: 24 Months
Population: EQ-5D score increase reported. 144 were analyzed as 10 patients were lost to follow-up and three were revised prior to a 24-month visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tornier Pyrocarbon Humeral Head
Number analyzed (Participants) | 144
units on a scale
  EQ-5D Increase (Change from baseline) | .21 (.15)
  EQ-5D (Absolute value) | .87 (.14)

6. Secondary Outcome: Pain Measured by a VIsual Analog Scale (VAS)
Description: Pain is measured by a visual analog scale (from 0-10). The subject responds to the question: How bad is your pain TODAY. 0 is no pain; 10 is pain as bad as it can be.
  Change in pain measured by a visual analog scale (VAS) at 24 months compared to baseline
Time Frame: 24 Months
Population: Change in Pain by VAS reported (decrease in pain). 144 were analyzed as 10 patients were lost to follow-up and three patients were revised prior to a 24-month visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tornier Pyrocarbon Humeral Head
Number analyzed (Participants) | 144
score on a scale
  Change in Pain by VAS reported (decrease in pain) | 4.23 (2.84)
  Pain by VAS (Absolute value) | 1.14 (1.88)

7. Secondary Outcome: Range of Motion (ROM)
Description: Range of Motion (ROM) is a movement test conducted on a joint to diagnose level of pain and function. The shoulder joint has a greater Range of Motion than all other joints in the body. In this study, ROM was measured using a goniometer for forward flexion in relation to the thorax, abduction, and external rotation (arm at side and arm abducted to 90°).
  Change in Range of Motion (ROM) at 24 months compared to baseline.
  * Forward Flexion
  * Abduction
  * External Rotation
Time Frame: 24 Months
Population: 144 patients were analyzed as 10 patients were lost to follow-up and three patients were revised prior to a 24-month visit.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Tornier Pyrocarbon Humeral Head
Number analyzed (Participants) | 144
Degrees
  Forward Flexion Increase | 33.5 (31.5)
  Abduction Increase | 43.5 (37.3)
  External Rotation Increase | 37.5 (28.6)

8. Secondary Outcome: Strength
Description: The subject's strength will be assessed using a fixed force gauge. The fixed force gauge is held in place by the examiner and the subject pulls upward with maximum effort for approximately five seconds. The test can be completed up to three times and the maximum score is used, however all three pulls will be recorded. The test is done only on the affected arm. The result of this test contributes to the Constant score calculation.
  Change in Strength testing at 24 months compared to baseline
Time Frame: 24 Months
Population: Increase in Strength reported. 144 were analyzed as 10 patients were lost to lost to follow-up and three patients were revised prior to a 24-month visit.
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Tornier Pyrocarbon Humeral Head
Number analyzed (Participants) | 144
Pounds
  Increase in Strength | 5 (7.6)
  Strength (Absolute value) | 14.8 (6.8)

9. Secondary Outcome: Number of Participants With Device-related Serious Adverse Events
Description: Adverse Events data will be collected and summarized at 24 months.
Time Frame: 24 Months
Population: Device-related Serious Adverse Events
Measure: Count of Participants; unit: Participants
Arm/Group | Tornier Pyrocarbon Humeral Head
Number analyzed (Participants) | 157
Participants | 5

10. Secondary Outcome: Revision Rate
Description: A revision is a procedure that adjusts or in any way modifies or removes any component of the original implant configuration, with or without replacement of a component, after the initial surgery. A revision may also include adjusting the position of the original configuration. An explant is a revision that includes permanent removal of any system component. If a subject has a revision that includes an addition of a glenoid component (revision to TSA) the Pyrocarbon humeral head must be permanently explanted.
  The Revision Rate will be calculated and summarized at 24 months.
Time Frame: 24 Months
Population: 147 were analyzed as 10 patients were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Tornier Pyrocarbon Humeral Head
Number analyzed (Participants) | 147
Participants | 3

11. Secondary Outcome: Level of Satisfaction With the Shoulder
Description: The level of satisfaction with the shoulder will be summarized at 24 months.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Groups:
- Tornier Pyrocarbon Humeral Head: The Tornier Pyrocarbon Humeral Head associated with the Tornier Flex stem.
Arm/Group | Tornier Pyrocarbon Humeral Head
Number analyzed (Participants) | 144
Participants
  Very Satisfied | 111
  Satisfied | 20
  Dissatisfied | 8
  Very Dissatisfied | 5

12. Secondary Outcome: X-Ray Data
Description: The follow data will be summarized at 24 Months:
  glenohumeral joint space width, glenoid osteophytes, glenoid morphology, humeral component radiolucency, osteolysis, migration, subsidence, subluxation, acromial humeral distance, anatomic fracture, and additional observations
Time Frame: 24 Months
Population: 144 subjects were analyzed as 10 subjects were lost to follow-up and three patients were revised prior to a 24-month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Tornier Pyrocarbon Humeral Head
Number analyzed (Participants) | 144
Participants
  Humeral Component Migration | 0
  Humeral Component Subsidence | 0
  Humeral Head Integrity | 0
  Glenoid Osteophytes Present | 78
  Humeral Component Radiolucency Present (< 1 mm) | 5
  Humeral Component Radiolucency Present (> 1 mm) | 0
  Humeral Component Osteolysis Present | 0
  Glenohumeral Subluxation Present (Slight) | 1
  Glenohumeral Subluxation Present (Moderate) | 0
  Anatomic Fracture (Present) | 1
  Glenohumeral Joint Space (< 3 mm) | 120
  Glenohumeral Joint Space (> 3 mm and < 6 mm) | 24
  Glenoid Morphology (None) | 25
  Glenoid Morphology (A1) | 58
  Glenoid Morphology (A2) | 40
  Glenoid Morphology (B1) | 4
  Glenoid Morphology (B2) | 14
  Glenoid Morphology (C) | 2
  Glenoid Morphology (Unable to assess) | 1
  Acromiohumeral Distance (> 2mm and < 7mm) | 31
  Acromiohumeral Distance (> 7mm) | 113

ADVERSE EVENTS:
Time Frame: Adverse events were collected from subject enrollment to the end of participation in the study which included two years of follow-up.
Description: An Adverse Event is any unfavorable or unintended sign, symptom, condition or disease in a study subject, where the experience occurs during the course of the study; regardless of its relationship to the test product or surgical procedure. For the purpose of this study, investigators are required to report all adverse events.
Arm/Group | Tornier Pyrocarbon Humeral Head
All-Cause Mortality (participants affected / at risk) | 0/157
Serious Adverse Events (participants affected / at risk) | 5/157
Other Adverse Events (participants affected / at risk) | 45/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tornier Pyrocarbon Humeral Head (N=157)
ARTHROFIBROSIS, TREATED SHOULDER (Musculoskeletal and connective tissue disorders) | 1 (1)
UNEXPECTED POSITIVE CULTURE (Musculoskeletal and connective tissue disorders) | 1 (1)
ROTATOR CUFF TEAR, TREATED SHOULDER (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN, TREATED SHOULDER; INFECTION, TREATED SHOULDER (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Treated Shoulder; MVC; Cervical Spondylosis (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tornier Pyrocarbon Humeral Head (N=157)
Pain, Treated Shoulder (Musculoskeletal and connective tissue disorders) | 21 (25)
Pain, Contralateral Shoulder (Musculoskeletal and connective tissue disorders) | 24 (24)
OA, in other non-study shoulder joints (Musculoskeletal and connective tissue disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a manuscript for the multi-center Publication has not been submitted within twelve (12) months of the conclusion (as defined in the Protocol), abandonment or termination of the Study, then the Researchers may Publish a subset of multi-center results of the Study. Sponsor personnel shall be acknowledged in accordance with customary scientific practice.

DOCUMENTS (2):
  • Study Protocol (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT02525783/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT02525783/SAP_001.pdf